CLINICAL TRIAL: NCT02771912
Title: Randomised Study of Propofol Versus Placebo for Sedation During Cataract Surgery Under Topical Anesthesia
Brief Title: Patient-controlled Sedation With Propofol During Cataract Surgery Under Topical Anesthesia
Acronym: CATARSIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILC_2016_5
Record Dates: First submitted 2016-05-12; First posted 2016-05-13 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Sedation
MeSH Terms: interventions — Propofol; soybean oil, phospholipid emulsion

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Propofol (Experimental): Infusion containing Propofol lipuro® 2% at a concentration of 2 mg/ml (100 ml of 5% glucose at which is removed 20 ml replaced with 20 ml of Propofol lipuro® 2 %).
  Self administration of propofol via patient-controlled sedation pump (ambIT pump) : bolus of 0.125 ml/kg of the solution (0.25 mg/kg propofol) with a programmed lock-out period of 3 minutes.
  Maximal dose of propofol : 1,25 mg/kg corresponding to 5mg/kg/h.
  Interventions: Drug: Propofol
- Intralipid (Placebo Comparator): Infusion containing Intralipid® (100 ml of 5% glucose at which is removed 20 ml replaced with 20 ml of Intralipid® 20%) to obtain an identical aspect to that of propofol infusion.
  Self administration via patient-controlled sedation pump (ambIT pump) : bolus of 0.125 ml/kg of the solution with a programmed lock-out period of 3 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propofol — Propofol and excipients
  Other Names: Propofol lipuro 2%
  Arms: Propofol
Drug: Placebo — Qualitative composition of Propofol lipuro 2% excipients
  Other Names: Intralipid
  Arms: Intralipid

SUMMARY:
Controversies exist about the use of propofol in sedation of patients for cataract surgery. This prospective randomised double-blind study evaluates the efficacy of patient-controlled sedation compared with placebo using the same device.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be operated of cataract under topical anesthesia

Exclusion Criteria:

* Contra-indication to sedation
* Complicated cataract
* Hypersensitivity to propofol, known or suspected hypersensitivity to egg phospholipid, soybean or peanut protein
* State of acute shock, severe dyslipidemia, severe liver failure, serious bleeding disorders
* Comprehension and language impairment
* Written and signed informed consent by the patient to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07; Primary Completion 2017-02-21 (Actual); Study Completion 2017-02-21 (Actual)

PRIMARY OUTCOMES:
Number of self administered bolus | One day

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmique Adolphe de Rothschild, Paris, France